CLINICAL TRIAL: NCT02518048
Title: A Phase 2a Trial Evaluating the Anti-psoriatic Effect of LEO 90100 Aerosol Foam Compared to Betesil® Medicated Plaster in the Treatment of Psoriasis Vulgaris
Brief Title: A Psoriasis Plaque Test Trial With LEO 90100 Compared to Betesil® in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0053-1227
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2017-05

CONDITIONS: Skin and Connective Tissue Diseases
Keywords: Psoriasis
MeSH Terms: conditions — Skin and Connective Tissue Diseases; Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 90100 Aerosol foam (Active Comparator): Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g (LEO 90100 Aerosol foam)
  Interventions: Drug: LEO 90100 Aerosol foam
- Betesil® 2.25 mg (Active Comparator): Betamethasone (as valerate). Each 7.5 cm x 10 cm medicated plaster contains: 2.250 mg of betamethasone valerate (corresponding to 1.845 mg of betamethasone).(Betesil® )
  Interventions: Drug: Betesil® 2.25 mg

INTERVENTIONS:
Drug: LEO 90100 Aerosol foam
  Arms: LEO 90100 Aerosol foam
Drug: Betesil® 2.25 mg
  Arms: Betesil® 2.25 mg

SUMMARY:
The purpose of this study is to evaluate the anti-psoriatic effect of LEO 90100 aerosol foam compared with Betesil® medicated plaster

DETAILED DESCRIPTION:
The products will be applied on 6 test sites (each product on 3 test sites) once daily 6 days a week (except Sundays) for 4 weeks. The application sites for each product will be determined according to random assignment. Depending on the size of the psoriasis plaques, 2 or 4 test sites will be located within the same plaque; the treatment assignment will be done pair-wise.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained
* Subjects with a diagnosis of psoriasis vulgaris with preferably three lesions (plaques) located on arms, legs and/or trunk or at least two lesions (plaques) located on arms, legs and/or trunk. For subjects with three lesions, each lesion must have a size suitable to accommodate 2 test sites (test site area 5 cm2, distance between two test sites at least 2 cm). For subjects with two lesions, one lesion must have a size suitable to accommodate 4 test sites, and the other lesion must accommodate 2 test sites.
* Age 18 years or above
* Outpatients
* Female subjects must be of either

  * non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus or has tubal ligation) or,
  * child-bearing potential provided there is a confirmed negative pregnancy test prior to trial treatment to rule out pregnancy.

Exclusion Criteria:

* Female subjects who are breast feeding
* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * Etanercept - within 4 weeks prior to randomisation and during the trial
  * Adalimumab, infliximab - within 8 weeks prior to randomisation and during the trial
  * Ustekinumab - within 16 weeks prior to randomisation and during the trial
  * Other products - within 4 weeks/5 half-lives prior to randomisation and during the trial (whichever is longer)
* Systemic treatment with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4-week period prior to randomisation and during the trial
* Subjects using phototherapy within the following time periods prior to randomisation and during the trial:

  * PUVA: 4 weeks
  * UVB: 2 weeks
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the trial:

  * Potent or very potent (WHO group III-IV) corticosteroids
* Subjects using one of the following topical drugs for the treatment of psoriasis within 2 weeks prior to randomisation and during the trial:

  * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis)
  * Topical retinoids, Vitamin D analogues, Topical immunomodulators (e.g. calcineurin inhibitors), Tar products, Salicylic acid
* Subjects using emollients on the selected plaques within 1 week before randomisation and during the trial
* Initiation of, or expected changes to concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, antimalarial drugs, lithium and ACE inhibitors) within 2 weeks prior to the randomisation and during the trial
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Queille-Roussel C, Rosen M, Clonier F, Norremark K, Lacour JP. Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Aerosol Foam Compared with Betamethasone 17-Valerate-Medicated Plaster for the Treatment of Psoriasis. Clin Drug Investig. 2017 Apr;37(4):355-361. doi: 10.1007/s40261-016-0489-5. PMID 27995521
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- LEO 90100 Aerosol Foam; Betesil® 2.25 mg: Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g (LEO 90100 Aerosol foam)
  LEO 90100 Aerosol foam
  Betamethasone (as valerate). Each 7.5 cm x 10 cm medicated plaster contains: 2.250 mg of betamethasone valerate (corresponding to 1.845 mg of betamethasone)
  Betesil® 2.25 mg
Period: Overall Study
Arm/Group | LEO 90100 Aerosol Foam; Betesil® 2.25 mg
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 35 subjects from 1 centre in France were enrolled into the trial. The first subject was enrolled on 22-Sep-2015 and the last subject completed the trial (last visit, including follow-up) on 07-Dec-2015.
Groups:
- All Study Participants: Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g (LEO 90100 Aerosol foam)
  LEO 90100 Aerosol foam
  Betamethasone (as valerate). Each 7.5 cm x 10 cm medicated plaster contains: 2.250 mg of betamethasone valerate (corresponding to 1.845 mg of betamethasone)
  Betesil® 2.25 mg
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25
Region of Enrollment [Number; unit: participants]
  France | 35

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Clinical Score (TCS) of Clinical Signs (Sum of Erythema, Scaling, Infiltration) Absolute Change in Total Clinical Score (TCS) of Clinical Signs (Sum of Erythema, Scaling, and Infiltration) at End of Treatment Compared to Baseline
Description: The investigator assessed the severity of the clinical signs erythema, scaling, and infiltration for each test site by using a 7-point scale with half-mark values from 0 (no evidence) to 3.0 (severe).
  The total TCS was calculated for each test site by summing the scores for erythema, scaling, and infiltration for that particular test site.
  Each test site was assessed at Baseline and on Days 4, 8, 11, 15, 18, 22, 25, and 29 (EoT).
  The mean TCS at Baseline was 6.6 for both groups.
Time Frame: Day 1 (Baseline) to Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LEO 90100 Aerosol Foam: Calcipotriol (as monohydrate) 50 mcg/g and betamethasone (as dipropionate) 0.5 mg/g (LEO 90100 Aerosol foam)
  LEO 90100 Aerosol foam
- Betesil® 2.25 mg: Betamethasone (as valerate). Each 7.5 cm x 10 cm medicated plaster contains: 2.250 mg of betamethasone valerate (corresponding to 1.845 mg of betamethasone)
  Betesil® 2.25 mg
Arm/Group | LEO 90100 Aerosol Foam | Betesil® 2.25 mg
Number analyzed (Participants) | 35 | 35
units on a scale
  TCS at Baseline | 6.6 (0.6) | 6.6 (0.6)
  Change in TCS Baseline to EoT | -5.8 (1.1) | -3.6 (1.5)
Statistical Analysis 1: Comparison: LEO 90100 Aerosol Foam vs Betesil® 2.25 mg; A last observation carried forward (LOCF) approach was used to account for drop-outs and missing values in the analysis of end of treatment values; Test type: Superiority or Other; p < 0.001, ANOVA — Least Square Means difference from ANOVA with treatment group as fixed effect and subject as random effect (105 treated sites per treatment group); Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-2.58 to -1.76]

2. Secondary Outcome: Change in TCS at Individual Visits
Time Frame: Day 1 (Baseline) to Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 90100 Aerosol Foam | Betesil® 2.25 mg
Number analyzed (Participants) | 35 | 35
units on a scale
  Day 4/Visit 5 | -1.3 (0.8) | -1.3 (0.7)
  Day 8/Visit 8 | -3.2 (1.2) | -2.0 (1.1)
  Day 11/Visit 11 | -4.3 (1.1) | -2.4 (1.4)
  Day 15/Visit 15 | -4.8 (1.2) | -2.8 (1.4)
  Day 18/Visit 18 | -5.1 (1.2) | -3.1 (1.5)
  Day 22/Visit 20 | -5.5 (1.2) | -3.2 (1.6)
  Day 25/Visit 23 | -5.7 (1.1) | -3.6 (1.6)
  Day 29/Visit 26 | -5.9 (1.1) | -3.7 (1.6)

3. Secondary Outcome: Change in Score of Erythema, Scaling, and Infiltration at Individual Visits
Description: The investigator assessed the severity of the clinical signs erythema, scaling, and infiltration for each test site by using a 7-point scale with half-mark values from 0 (no evidence) to 3.0 (severe).
  Erythema: 0 (no evidence - normal skin color) to 3 (severe - intense red). Scaling: 0 (no evidence - no scaling) to 3 (severe - coarse, thick scales). Infiltration: 0 (no evidence - no infiltration) to 3 (severe - very marked infiltration).
Time Frame: Day 1 (Baseline) to Day 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 90100 Aerosol Foam | Betesil® 2.25 mg
Number analyzed (Participants) | 35 | 35
units on a scale
  Erythema Day 4/Visit 5 | -0.5 (0.4) | -0.4 (0.4)
  Erythema Day 8/Visit 8 | -0.9 (0.4) | -0.6 (0.4)
  Erythema Day 11/Visit 11 | -1.3 (0.5) | -0.8 (0.5)
  Erythema Day 15/Visit 14 | -1.4 (0.5) | -0.9 (0.5)
  Erythema Day 18/Visit 17 | -1.6 (0.6) | -1.0 (0.6)
  Erythema Day 22/Visit 20 | -1.7 (0.6) | -1.1 (0.6)
  Erythema Day 25/Visit 23 | -1.8 (0.6) | -1.3 (0.6)
  Erythema Day 29/Visit 26 | -1.9 (0.5) | -1.2 (0.6)
  Scaling Day 4/Visit 5 | -0.6 (0.3) | -0.6 (0.3)
  Scaling Day 8/Visit 8 | -1.3 (0.5) | -0.8 (0.5)
  Scaling Day 11/Visit 11 | -1.7 (0.5) | -1.0 (0.6)
  Scaling Day 15/Visit 14 | -1.8 (0.5) | -1.1 (0.6)
  Scaling Day 18/Visit 17 | -1.9 (0.5) | -1.2 (0.6)
  Scaling Day 22/Visit 20 | -2.0 (0.5) | -1.2 (0.6)
  Scaling Day 25/Visit 23 | -2.0 (0.4) | -1.4 (0.6)
  Scaling Day 29/Visit 26 | -2.0 (0.4) | -1.3 (0.6)
  Infiltration Day 4/Visit 5 | -0.3 (0.2) | -0.3 (0.2)
  Infiltration Day 8/Visit 8 | -0.9 (0.5) | -0.5 (0.4)
  Infiltration Day 11/Visit 11 | -1.3 (0.4) | -0.6 (0.5)
  Infiltration Day 15/Visit 14 | -1.6 (0.4) | -0.8 (0.5)
  Infiltration Day 18/Visit 17 | -1.7 (0.4) | -0.8 (0.6)
  Infiltration Day 22/Visit 20 | -1.8 (0.3) | -0.9 (0.6)
  Infiltration Day 25/Visit 23 | -1.9 (0.3) | -1.0 (0.6)
  Infiltration Day 29/Visit 26 | -1.9 (0.3) | -1.1 (0.6)

4. Secondary Outcome: Change in Total Skin Thickness and Echo-poor Band Thickness From Baseline to EoT
Description: Skin thickness ultrasound measurements of the test sites were performed at Baseline and End of Treatment.
  Two skin parameters were calculated using ultrasound:
  * The mean total skin thickness
  * The mean echo-poor band thickness
Time Frame: Baseline to End of Treatment
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | LEO 90100 Aerosol Foam | Betesil® 2.25 mg
Number analyzed (Participants) | 35 | 35
millimeters
  Change in Total Skin Thickness | -1.0 (0.3) | -0.6 (0.4)
  Change in Echo-Poor Band Thickness | -1.3 (0.5) | -0.7 (0.5)
Statistical Analysis 1: Comparison: LEO 90100 Aerosol Foam vs Betesil® 2.25 mg; Total Skin Thickness: LEO 90100 vs. Betesil®; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.53 to -0.32]
Statistical Analysis 2: Comparison: LEO 90100 Aerosol Foam vs Betesil® 2.25 mg; Echo-Poor Band Thickness: LEO 90100 vs. Betesil®; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.69 to -0.41]

ADVERSE EVENTS:
Time Frame: From signed Informed consent form (Day -28 to -1) to end of Follow-up (Day 43 +/-2).
Groups:
- All Subjects: All subjects received both medication and reporting is on the entire population.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 15/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=35)
Headache (Nervous system disorders) | 5 (8)
Influenza (Infections and infestations) | 3 (3)
Hordeolum (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before submitting or presenting a manuscript about the clinical trial to a third party, the investigator shall give LEO a copy of any such manuscript, and LEO has the right to review and comment. Upon the request of LEO, the investigator shall remove any confidential information before submitting or presenting a manuscript. To allow LEO to protect its inventions and other intellectual property rights, the publication or presentation can be delayed.